CLINICAL TRIAL: NCT03976973
Title: A Phase 2, Multi-centre Study of BromAc for Recurrent Peritoneal Mucinous Tumour or Pseudomyxoma Peritonei
Brief Title: BromAc for Recurrent Peritoneal Mucinous Tumour or Pseudomyxoma Peritonei
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mucpharm Pty Ltd (Industry)
Collaborators: Mercy Medical Center (Other); Wake Forest University Health Sciences (Other); University of Pittsburgh Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUC-ONC-ACP2
Record Dates: First submitted 2019-05-24; First posted 2019-06-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Pseudomyxoma Peritonei; Peritoneal Cancer; Mucinous Adenocarcinoma; Mucinous Tumor
MeSH Terms: conditions — Pseudomyxoma Peritonei; Adenocarcinoma, Mucinous; Neoplasms, Cystic, Mucinous, and Serous | interventions — Bromelains; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants with inoperable pseudomyxoma peritonei or peritoneal mucinous tumour that meet the entry criteria and consent to the intervention will receive intratumoural treatment/s with the combination drug BromAc. The drug product will be injected directly into the tumour via a radiologically placed drain
  Interventions: Drug: Bromelain; Drug: Acetylcysteine; Procedure: Interventional radiology insertion of drain

INTERVENTIONS:
Drug: Bromelain — Intratumoural injections of Bromelain 600ug/ml (maximum dose 90mg daily diluted in 150ml 0.9% NaCl) via a radiologically placed drain in combination with Acetylcysteine in 0.9% sodium chloride (normal saline).
Drug: Acetylcysteine — Intratumoural injections of Acetylcysteine 20mg/ml (maximum dose 3g daily diluted in 150ml 0.9% NaCl) via a radiologically placed drain in combination with Bromelain.
Procedure: Interventional radiology insertion of drain — Under radiological guidance (CT), a needle, wire, dilator will be placed directly into the tumour, then a pigtail drain (10Frg) will be secured into the tumour by an experienced, interventional radiologist, under standard procedures. This drain is utilised as access to the tumour for injections of the investigational drug product BromAc, and subsequent aspirations.

SUMMARY:
Pseudomyxoma peritonei (PMP) is an orphan disease, characterized by the progressive accumulation of jelly-like material within the abdomen, which occurs in approximately 2-3 people per million per year. Advanced disease is often the result of tumour perforation and seeding of tumour cells within the peritoneal cavity. Complete cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CCRS HIPEC) is the current standard of care for PMP.

An Australian pharmaceutical company is developing BromAc for diseases involving mucin. This drug is composed of Bromelain and Acetylcysteine. During pre-clinical development, the sponsor found that BromAc rapidly dissolved and removed tumour mucin, making it a potent mucolytic. BromAc in combination have the ability, as shown in pre-clinical studies, to remove the mucin protective framework expressed by cancer including mucin (MUC) 1, MUC2, MUC4, MUC5AC and MUC16. The sponsor has shown the mechanism of action of BromAc - to break peptide and glycosidic linkages and disulphide bonds in tumour produced and respiratory mucin. BromAc has been safe in preclinical development with a manageable adverse event profile and preliminary efficacy in a phase 1 study.

This current study will examine the efficacy and safety of applying BromAc directly into recurrent mucinous tumour deposits in patients that are found to be unsuitable for repeat curative intent intervention by CCRS HIPEC.

DETAILED DESCRIPTION:
Pseudomyxoma peritonei (PMP) is an orphan disease, characterised by the progressive accumulation of jelly-like material within the abdomen, which occurs in approximately 3 people per million per year. Advanced disease is often the result of tumour perforation and seeding of tumour cells within the peritoneal cavity, leading to this syndrome. Multifocal mucin collections are the main cause of morbidity and mortality.

In the past, management of mucinous peritoneal disease involved repeated surgical debulking, with systemic chemotherapy having minimal effect. The combined modality of complete cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CCRS HIPEC) is considered standard of care for peritoneal spread of appendiceal tumours and a treatment option for other mucinous peritoneal tumours. The intention of CCRS HIPEC is cure, however this is dependent on the characteristics and extent of tumour involvement, with the main limitation being amount of disease involving the serosa or mesentery of small bowel.

Mucin produced by tumours is known to be highly resistant to chemotherapy as mucin acts as a tumour coating. Many patients with mucinous tumours or PMP, however, can achieve long-term survival through this therapy although in a significant proportion recurrence following CCRS HIPEC occurs, and repeat interventions for recurrent disease are increasingly complex and may have a negative impact on quality of life, where the risks of the procedure in many cases outweigh the benefits.

BromAc has been safe in preclinical development and in a phase 1 study, patients received up to 60mg/2000mg of BromAc daily for a median of 3.4 days. Serious treatment-related adverse events (12%) were manageable. There were no anaphylactic reactions. An objective response to treatment was seen in 81% of patients. There were no drug-related deaths due to treatment-related adverse events. With a median follow up of 18.2 months, progression was seen in 55% at a median of 5.8 months.

This potential treatment for pseudomyxoma peritonei/appendix mucinous tumours received orphan designation from the (Food and Drug Administration (FDA) (DRU-2018-6644) European Medicines Agency (EMA) (EMA/3/18/2107, EMA/3/18/2113).

The aim of this study is to assess whether the application of BromAc via radiologically placed percutaneous catheters directly into the recurrence dissolves the mucinous tumour, allowing for the dissolved tumour to be drained. The efficacy of this intervention will be assessed via radiological imaging and clinically with the expectation that this combination treatment will result in dissolution and removal of the tumour. The surrogate endpoints used in this study will be radiological response and volume of mucin aspirated. The projected benefits of direct injection of the BromAc include improvement of symptoms of the disease, which frequently include pain, vomiting, inability to maintain adequate oral intake and progressive loss of condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 80 years
* Have a mucinous tumour/pseudomyxoma peritonei target lesion with a defined cavity, with the shortest diameter being at least 3 centimeters on radiology, and percutaneously accessible. In the case of a target lesion, tumour located at distant sites (for e.g. pleura) will not exclude a patient from this study and these tumours may be treated, if suitable, under expanded access protocols.
* Are symptomatic or at risk of becoming symptomatic or obstructed imminently, are considered inoperable, at high risk of morbidity, mortality or quality of life decline for repeat surgery, or do not wish to explore repeat surgery
* Are considered suitable for the trial based on a multidisciplinary team meeting case review

Exclusion Criteria:

* Have a non-mucinous tumour (hard caked tumour) that does not have cystic appearance on radiology. Having a hard tumour appearance in one region does not exclude treatment in another area, provided the appearance is mucinous.
* Have suspected fistula of the tumour into the gastrointestinal tract, invading or abutting major vessel or other area of concern (fistulation into bladder or vaginal cuff is not an exclusion for treatment)
* Have known allergy (anaphylaxis) or allergy to pineapples, papain, bromeliads, sulphur, eggs or Acetylcysteine or any other serious allergy or intolerance to fruits or food products
* Have a coagulation disorder of any kind or are on anticoagulant or anti-platelet therapy that cannot be managed or withheld for the radiology procedure
* Have an infected tumour or ongoing inflammatory process (pus on aspiration at radiology will be a delayed failure) as indicated on baseline blood test
* Eastern Cooperative Oncology Group (ECOG) score >2
* Have had chemotherapy within the last two weeks, have not had bone marrow recovery from chemotherapy, or had Bevacizumab (Avastin) within the last 4 weeks. A staging baseline scan must be completed prior to considering entry into this study.
* Have previously received BromAc for pseudomyxoma or peritoneal mucinous tumour (see expanded access)
* Have other serious comorbidities where inclusion in the trial will subject the participant to an unacceptable higher risk of adverse events as judged by the investigator
* Pregnant women are excluded from this study because BromAc has unknown but a potential risk for adverse events in nursing infants secondary to treatment of the mother
* Participants with psychiatric illness/social situations that would limit compliance with study requirements
* Are unable to give fully informed and educated consent or are unable to comply with the standard follow up procedures of a clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Tumour response (objective response rate) | 1 month
  Tumour changes following BromAc combination treatment compared to baseline. Efficacy will be measured by RECIST v1.1 with the volume of fluid aspirated from the drain (dissolved tumour). The treatment will be seen effective if >30% of tumour volume is aspirated or there is a >30% reduction on CT scan post treatment at 1 month compared to the pre-treatment scan. Given the difficulty of assessing soft tumour (cystic/mucinous) response by RECIST, a surrogate assessment of efficacy will be measured (if unable to assess based on RECIST v1.1 criteria) by tumour changes following BromAc combination treatment.

SECONDARY OUTCOMES:
Progression free survival post treatment | 1 month, 3 months, 6 months, 9 months and 12 months
  Time to progression of the treated area (duration of response) based on repeat CT scanning where RECIST v1.1 will be used where possible. The follow up scan will be compared to the 1 month post treatment scan where dimensions and volume will be calculated by an experienced radiologist.
Impact of treatment on Quality of Life over time in patients evaluated by the core questionnaire 'European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Cancer (EORTC-QLQ-C30)'. | Baseline, then at 1 month, 3 months, 6 months, 9 months and 12 months
  The EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Core - C30) is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items.
  The global health status / Quality of Life scale has scores from 1 (very poor) to 7 (excellent) and the others from 1 (not at all) to 4 (very much) where 4 is the worst score. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Impact of treatment on Quality of Life in colorectal cancer over time by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Colorectal Cancers (EORTC-QLQ-CR29) | Baseline, then at 1 month, 3 months, 6 months, 9 months and 12 months
  The symptom scores (Fatigue, Nausea and vomiting, Pain …), with scores from 1 (not at all) to 4 (very much), where 4 is the worst score, will be evaluated by the use of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Colorectal Cancer (EORTC-QLQ-CR29). The trend of each category of outcome measures given by the EORTC-QLQ-CR29 in four groups of patients: tumour on the right and transverse part of the colon; tumour on the left part of the colon; rectal tumour; metastatic colorectal cancer.
Incidence of Treatment-Emergent Adverse Events (Pathology) [Safety and Tolerability] | 1 month
  Reported as any untoward medical occurrence or worsening of a pre-existing medical condition in a participant administered BromAc, and judged possibly, probably, or definitely related to treatment
Symptomatic response to treatment | Baseline, 1 week, 1 month, 3 months, 6 months, 9 months and 12 months
  Symptoms from tumour will be assessed at baseline then compared to post treatment symptoms to determine resolution or worsening of symptoms from tumour experienced.
Laboratory blood test parameters | Baseline, 1 week, 1 month, 3 months, 6 months, 9 months and 12 months
  Laboratory parameters (haematology, clinical chemistry and coagulation) will be assessed at baseline then at each interval to assess for any alteration compared to baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Armando Sardi, MD, Principal Investigator — Mercy Medical Center, USA; Haroon Choudry, MD, Principal Investigator — University of Pittsburgh Medical Center, USA; Edward Levine, MD, Principal Investigator — Wake Forest University Hospital, USA; Alvaro Arjona Sanchez, MD, Principal Investigator — University Hospital Reina Sofia, Spain; Ignace de Hingh, MD, Principal Investigator — Eindhoven Catharina Hospital, Netherlands

IPD SHARING:
Plan to Share IPD: No